CLINICAL TRIAL: NCT03412565
Title: A Multicenter Phase 2 Study to Evaluate Subcutaneous Daratumumab in Combination With Standard Multiple Myeloma Treatment Regimens
Brief Title: A Study to Evaluate Subcutaneous Daratumumab in Combination With Standard Multiple Myeloma Treatment Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108435; 2017-004203-41 (EudraCT Number); 54767414MMY2040 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone; Melphalan; Prednisone; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Daratumumab(D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) (Experimental): Participants will receive daratumumab 1800 milligram (mg) by subcutaneous (SC) injection on Days 1, 8 and 15 of Cycles 1 to 3 (each cycle of 21 days) and on Day 1 of Cycle 4; bortezomib 1.3 milligram per square meter (mg/m^2) SC injection on Days 1, 4, 8 and 11 of Cycles 1 to 4; lenalidomide 25 mg orally on Day 1 through Day 14 of Cycles 1 to 4 and dexamethasone 20 mg orally or intravenously on Days 1, 2 ,8, 9, 15 and 16 of Cycle 1 to 4.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- D + Bortezomib + Melphalan + Prednisone (D-VMP) (Experimental): Participants will receive daratumumab 1800 mg by SC injection on Days 1, 8, 15, 22, 29 and 36 of Cycle 1 then on Days 1 and 22 in Cycles 2 to 9 and Day 1 of Cycle 10 and thereafter until documented progression of disease, unacceptable toxicity, or end of study; bortezomib 1.3 mg/m^2 SC injection on Day 1, 4, 8, 11, 22, 25, 29 and 32 of Cycle 1 and on Days 1, 8, 22 and 29 of Cycles 2 to 9; melphalan 9 mg/m^2 orally on Day 1 through Day 4 of Cycles 1 to 9; prednisone 60 mg/m^2 orally on Days 1 to 4 of cycles 1 to 9.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Melphalan; Drug: Prednisone
- Daratumumab + Lenalidomide + Dexamethasone (D-Rd) (Experimental): Participants will receive daratumumab 1800 mg by SC injection on Days 1, 8, 15 and 22 of Cycles 1 and 2 then on Day 1 and 15 of Cycles 3 to 6 and on Day 1 of Cycle 7 and thereafter until documented progression of disease, unacceptable toxicity, or end of study; lenalidomide 25 mg orally on Day 1 through Day 21 of each cycle until documented progression of disease, unacceptable toxicity, or end of study and dexamethasone 40 mg orally or intravenously weekly until documented progression of disease, unacceptable toxicity, or end of study.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone
- Daratumumab + Carfilzomib + Dexamethasone (D-Kd) (Experimental): Participants will receive daratumumab 1800 mg by SC injection on Days 1, 8, 15 and 22 of Cycles 1 and 2 (each cycle is of 28 days) then on Day 1 and 15 of Cycles 3 to 6 and on Day 1 of Cycle 7 and thereafter until documented progression of disease, unacceptable toxicity, or end of study; Carfilzomib 20 mg/m^2 intravenously (IV) on Day 1 of Cycle 1 only then 70 mg/m^2 IV on Days 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2 and thereafter until documented progression of disease, unacceptable toxicity, or end of study and dexamethasone 40 mg orally or IV weekly for Cycles 1-9 then on Days 1, 8, 15 of each cycle for Cycles 10 and thereafter until documented progression of disease, unacceptable toxicity, or end of study.
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered at a dose of 1800 mg by SC injection in Cycles 1 to 4 in D-VRd cohort and until documented progression of disease, unacceptable toxicity, or end of study for D-VMP, D-Rd and D-Kd cohorts.
Drug: Bortezomib — Bortezomib will be administered as 1.3 mg/m^2 SC injection in Cycles 1 to 4 in D-VRd cohort and in Cycles 1 to 9 in D-VMP cohort.
  Arms: D + Bortezomib + Melphalan + Prednisone (D-VMP); Daratumumab(D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd)
Drug: Lenalidomide — Lenalidomide will be administered as 25 mg capsule orally in Cycles 1 to 4 in D-VRd cohort and in all Cycles until documented progression of disease, unacceptable toxicity, or end of study in D-Rd cohort.
  Arms: Daratumumab + Lenalidomide + Dexamethasone (D-Rd); Daratumumab(D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd)
Drug: Dexamethasone — Dexamethasone will be administered as 20 mg orally or intravenously in Cycles 1 to 4 in D-VRd cohort; 40 mg orally or intravenously in all cycles and thereafter until documented progression of disease, unacceptable toxicity, or end of study in D-Rd and D-Kd cohort.
  Arms: Daratumumab + Carfilzomib + Dexamethasone (D-Kd); Daratumumab + Lenalidomide + Dexamethasone (D-Rd); Daratumumab(D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd)
Drug: Melphalan — Melphalan will be administered as 9 mg/m^2 orally in Cycles 1 to 9.
  Arms: D + Bortezomib + Melphalan + Prednisone (D-VMP)
Drug: Prednisone — Prednisone will be administered as 60 mg/m^2 orally in cycles 1 to 9.
  Arms: D + Bortezomib + Melphalan + Prednisone (D-VMP)
Drug: Carfilzomib — Carfilzomib will be administered as 20 mg/m^2 IV on Day 1 of Cycle 1 only then 70 mg/m^2 IV on Days 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2 and thereafter until documented progression of disease, unacceptable toxicity, or end of study in D-Kd cohort.
  Arms: Daratumumab + Carfilzomib + Dexamethasone (D-Kd)

SUMMARY:
The purpose of this study is to evaluate the clinical benefit of subcutaneous (SC) daratumumab administered in combination with standard multiple myeloma (MM) regimens in participants with MM as measured by overall response rate (ORR) or very good partial response (VGPR) or better rate.

DETAILED DESCRIPTION:
The hypothesis is that the addition of daratumumab administered SC to standard MM regimens will improve responses compared to response data observed in completed phase 3 studies without daratumumab. Disease evaluations will include measurements of myeloma proteins, bone marrow examinations, skeletal surveys, assessment of extramedullary plasmacytomas, and measurements of serum calcium corrected for albumin. Safety will be measured by adverse events, laboratory test results, electrocardiogram (ECGs), vital sign measurements, physical examination findings, SC injection-site assessments, and assessment of Eastern Cooperative Oncology Group (ECOG) performance status score. Study will consist of 3 phases (screening, treatment and follow-up) and duration of study is approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma diagnosed according to the International Myeloma Working Group (IMWG) diagnostic criteria
* Measurable, secretory disease as defined by any of the following:

  1. Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=) 1.0 gram per deciliter (g/dL); or
  2. Urine M-protein level >= 200 milligram per 24 hours (mg/24 hours); or
  3. Light chain multiple myeloma (MM), for participants without measurable disease in the serum or urine: serum Immunoglobulin (Ig) free light chain (FLC) >= 10 mg/dL and abnormal FLC ratio
* Meets one of the sets of the following criteria:

  1. For Daratumumab + bortezomib + lenalidomide + dexamethasone (D-VRd) and Daratumumab + bortezomib + melphalan + prednisone + dexamethasone (D-VMP) regimen: newly diagnosed myeloma
  2. For Daratumumab + lenalidomide + dexamethasone (D-Rd) and Daratumumab + Carfilzomib + Dexamethasone (D-Kd) regimen: relapsed or refractory disease
  3. D-Kd cohort: Participants must have received only 1 prior line of therapy for MM which included at least 2 consecutive cycles of lenalidomide therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0, 1, or 2
* During the study, during dose interruptions, and for 3 months after receiving the last dose of any component of the study treatment, a female participant must agree not to donate eggs (ova, oocytes) and male participants of reproductive potential must not donate semen or sperm during the study, during dose interruptions, or for 3 months after the last dose of any study drug

Exclusion Criteria:

* History of malignancy (other than MM) unless all treatment of that malignancy was completed at least 2 years before consent and the participant has no evidence of disease further exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or breast, or other non-invasive lesion, that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years
* Exhibits clinical signs of meningeal involvement of MM
* Either of the following: a) Chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) is less than (<) 50 percentage (%) of predicted normal b) Moderate or severe persistent asthma, or a history of asthma within the last 2 years, or currently has uncontrolled asthma of any classification c) For D-Kd cohort: Known infiltrative pulmonary disease or known pulmonary hypertension
* Any of the following: a) Known to be seropositive for human immunodeficiency virus; b) Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [Anti-HBc] and/or antibodies to hepatitis B surface antigen [Anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are polymerase chain reaction (PCR) positive will be excluded
* Known to be seropositive for hepatitis C (Anti-HCV antibody positive or HCV-RNA quantitation positive) except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy
* For D-Kd cohort only: Transthoracic echocardiogram showing left ventricular ejection fraction (LVEF) <40%; uncontrolled hypertension, defined as an average systolic blood pressure greater than (>)159 millimeters of mercury (mmHg) or diastolic >99 mmHg despite optimal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (64):
- United States (16):
  - Cancer Center of Central Connecticut - Southington, Southington, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Karmonos Cancer Institute, Detroit, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - Billings Clinic, Billings, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - San Juan Oncology Associates, Farmington, New Mexico
  - NYU Winthrop, Mineola, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Wake Forest University Baptist Medical Center (WFUBMC) - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Avera Medical Group - Oncology & Hematology, Sioux Falls, South Dakota
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Cancer Center - Emily Couric Clinical Cancer Center - Women's Oncology Clinic, Charlottesville, Virginia
- Brazil (6):
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo - Hospital Sao Vicente de Paulo, Passo Fundo
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Clinica Sao Germano, São Paulo
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze - I. interni klinika - klinika hematologie, Prague
- France (5):
  - CHU de Nantes hotel Dieu, Nantes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU Bretonneau, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Tuebingen der Eberhard-Karls-Universitaet, Abteilung fuer Innere Medizin II,, Tübingen
- Israel (6):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (4):
  - Kanazawa University Hospital, Kanazawa
  - Matsuyama Red Cross Hospital, Matsuyama
  - Nagoya City University Hospital, Nagoya
  - Japanese Red Cross Medical Center, Shibuya City
- Spain (12):
  - Inst. Cat. D'Oncologia-Badalona, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Son Llatzer, Mallorca
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Dr. Peset, Valencia
- United Kingdom (6):
  - Heart of England NHS Foundation Trust, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Kent and Canterbury Hospital, Canterbury
  - Manchester Royal Infirmary, Manchester
  - Derriford Hospital, Plymouth
  - Royal Stoke University Hospital, Stoke-on-Trent

REFERENCES:
- [Derived] Moreau P, Chari A, Oriol A, Martinez-Lopez J, Haenel M, Touzeau C, Ailawadhi S, Besemer B, de la Rubia Comos J, Encinas C, Mateos MV, Salwender H, Rodriguez-Otero P, Hulin C, Karlin L, Sureda Balari A, Bargay J, Benboubker L, Rosinol L, Tarantolo S, Terebelo H, Yang S, Wang J, Nnane I, Qi M, Kosh M, Delioukina M, Goldschmidt H. Daratumumab, carfilzomib, and dexamethasone in relapsed or refractory myeloma: final analysis of PLEIADES and EQUULEUS. Blood Cancer J. 2023 Mar 7;13(1):33. doi: 10.1038/s41408-023-00805-x. No abstract available. PMID 36882409

RESULTS

PARTICIPANT FLOW:
Groups:
- Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd): Participants received daratumumab 1800 milligrams (mg) as a subcutaneous (SC) injection on Days 1, 8 and 15 of Cycles 1 to 3 (each cycle of 21 days) and on Day 1 of Cycle 4; bortezomib 1.3 milligrams per square meter (mg/m^2) SC injection on Days 1, 4, 8 and 11 of Cycles 1 to 4; lenalidomide 25 mg orally on Day 1 through Day 14 of Cycles 1 to 4 and dexamethasone 20 mg orally or intravenously (IV) on Days 1, 2 ,8, 9, 15 and 16 of Cycle 1 to 4.
- D + Bortezomib + Melphalan + Prednisone (D-VMP): Participants received daratumumab 1800 mg by SC injection on Days 1, 8, 15, 22, 29 and 36 of Cycle 1, then on Days 1 and 22 in Cycles 2 to 9, and Day 1 of Cycle 10 and thereafter until documented progression of disease, unacceptable toxicity, or up to 2 years and 7 months; bortezomib 1.3 mg/m^2 SC injection on Day 1, 4, 8, 11, 22, 25, 29 and 32 of Cycle 1 and on Days 1, 8, 22 and 29 of Cycles 2 to 9; melphalan 9 mg/m^2 orally on Day 1 through Day 4 of Cycles 1 to 9; prednisone 60 mg/m^2 orally on Days 1 to 4 of cycles 1 to 9.
- Daratumumab + Lenalidomide + Dexamethasone (D-Rd): Participants received daratumumab 1800 mg by SC injection on Days 1, 8, 15 and 22 of Cycles 1 and 2, then on Day 1 and 15 of Cycles 3 to 6, and on Day 1 of Cycle 7 and thereafter until documented progression of disease, unacceptable toxicity, or up to 2 years and 7 months; lenalidomide 25 mg orally on Day 1 through Day 21 of each cycle until documented progression of disease, unacceptable toxicity, or end of study and dexamethasone 40 mg orally or intravenously weekly until documented progression of disease, unacceptable toxicity, or up to 2 years and 7 months.
- Daratumumab + Carfilzomib + Dexamethasone (D-Kd): Participants received daratumumab 1800 mg by SC injection on Days 1, 8, 15 and 22 of Cycles 1 and 2 (each cycle is of 28 days), then on Day 1 and 15 of Cycles 3 to 6, and on Day 1 of Cycle 7 and thereafter until documented progression of disease, unacceptable toxicity, or up to 2 years and 7 months; Carfilzomib 20 mg/m^2 IV on Day 1 of Cycle 1 only, then 70 mg/m^2 IV on Days 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2 and thereafter until documented progression of disease, unacceptable toxicity, or up to 2 years and 7 months and dexamethasone 40 mg orally or IV weekly for Cycles 1-9, then on Days 1, 8, 15 of each cycle for Cycle 10 and thereafter until documented progression of disease, unacceptable toxicity, or up to 2 years and 7 months.
Period: Overall Study
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Started | 67 | 67 | 65 | 66
Completed | 66 | 19 | 14 | 15
Not Completed | 1 | 48 | 51 | 51
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 5 | 5
Not completed — Death | 1 | 3 | 4 | 5
Not completed — Data collection ended | 0 | 41 | 41 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd) | Total
Number analyzed (Participants) | 67 | 67 | 65 | 66 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.47) | 74.9 (4.54) | 66.8 (9.58) | 61 (9.77) | 65 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 36 | 20 | 32 | 107
  Male | 48 | 31 | 45 | 34 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 0 | 7 | 16
  Not Hispanic or Latino | 34 | 39 | 45 | 43 | 161
  Unknown or Not Reported | 30 | 22 | 20 | 16 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 2 | 2 | 10
  White | 38 | 46 | 45 | 48 | 177
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 24 | 15 | 18 | 16 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 1 | 4 | 0 | 0 | 5
  CZECH REPUBLIC | 4 | 4 | 15 | 0 | 23
  FRANCE | 26 | 21 | 17 | 15 | 79
  GERMANY | 0 | 0 | 0 | 19 | 19
  ISRAEL | 0 | 7 | 14 | 0 | 21
  JAPAN | 0 | 4 | 0 | 0 | 4
  SPAIN | 11 | 19 | 0 | 25 | 55
  UNITED KINGDOM | 9 | 8 | 12 | 0 | 29
  UNITED STATES | 16 | 0 | 7 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: D-VMP, D-Rd, and D-Kd Cohorts: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved partial response (PR) or better according to international myeloma working group (IMWG) criteria. IMWG criteria for PR: greater than or equal to (>=) 50 percent (%) reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to less than (<) 200 milligrams (mg) per 24 hours, If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow plasma cells (PCs) is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Up to 2 years 3 months
Population: All treated analysis set included all participants who have received at least 1 dose of study treatment. This primary outcome measure (OM) was planned to be analyzed for D-VMP, D-Rd and D-Kd cohorts only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 67 | 65 | 66
percentage of participants | 88.1 [79.5 to 93.9] | 90.8 [82.6 to 95.9] | 84.8 [75.7 to 91.5]

2. Primary Outcome: D-VRd Cohort: Percentage of Participants With Very Good Partial Response (VGPR) or Better Response
Description: VGPR or better rate was defined as the percentage of participants who achieved VGPR or complete response (CR) (including stringent complete response [sCR]) according to the IMWG criteria during or after the study treatment. VGPR: Serum and urine component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein level <100 mg/24 hour; CR: negative immunofixation on the serum and urine, Disappearance of any soft tissue plasmacytomas and <5% PCs in bone marrow; sCR: CR in addition to having a normal FLC ratio and an absence of clonal cells in bone marrow by immunohistochemistry, immunofluorescence, 2-4 color flow cytometry.
Time Frame: Up to 2 years and 3 months
Population: All treated analysis set included all participants who have received at least 1 dose of study treatment. This primary outcome measure (OM) was planned to be analyzed for D-VRd cohort only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd)
Number analyzed (Participants) | 67
percentage of participants | 71.6 [61.2 to 80.6]

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Daratumumab
Description: Cmax was defined as maximum serum concentration observed following daratumumab administration. Each cycle for: D-VRd cohort is of 21 days, D-VMP cohort is of 42 days and D-Rd and D-Kd cohorts is of 28 days. Each cohort have a treatment period of 84 days.
Time Frame: D-VRd: Day 4 of Cycles 1 and 4 and post treatment at Week 8; D-VMP: Day 4 of Cycles 1 and 2 and post treatment at Week 8; D-Rd and D-Kd: Day 4 of Cycles 1 and 3 and post treatment at Week 8
Population: Pharmacokinetics (PK) analysis set: participants who received at least 1 dose of daratumumab SC and had at least 1 PK sample value after first dose. 'N' (number of participants analyzed): participants evaluated for this OM; 'n' (number analyzed): participants analyzed at specific timepoints. The "0" in the number analyzed field indicates that no participant was evaluable for PK at that timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 60 | 66 | 56 | 57
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 4 | 100 (48.5) | 98.6 (51.6) | 108 (49.9) | 137 (56.7)
  Cycle 2 Day 4: number analyzed (Participants) | 0 | 55 | 0 | 0
  Cycle 2 Day 4 |  | 612 (256) |  |
  Cycle 3 Day 4: number analyzed (Participants) | 0 | 0 | 50 | 45
  Cycle 3 Day 4 |  |  | 648 (238) | 869 (274)
  Cycle 4 Day 4: number analyzed (Participants) | 56 | 0 | 0 | 0
  Cycle 4 Day 4 | 746 (275) |  |  |
  Post-treatment Phase Week 8: number analyzed (Participants) | 43 | 1 | 0 | 6
  Post-treatment Phase Week 8 | 263 (190) | 162 (NA) — Standard deviation (SD) data is 0 as SD cannot be calculated for 1 participant. |  | 49.3 (109)

4. Secondary Outcome: Percentage of Participants With Infusion-Related Reactions (IRRs)
Description: Percentage of Participants with IRRs were reported. The administration-related systemic reactions are referred to as IRRs.
Time Frame: For D-VRD Arm: Baseline up to 2 years 3 months; For D-VMP, D-Rd and D-Kd Arms: Baseline up to 2 years 7 months
Population: All treated analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 67 | 67 | 65 | 66
percentage of participants | 9.0 [4.0 to 16.9] | 9.0 [4.0 to 16.9] | 4.6 [1.3 to 11.5] | 4.5 [1.3 to 11.3]

5. Secondary Outcome: D-VMP, D-Rd, and D-Kd Cohorts: Percentage of Participants With VGPR or Better Response
Description: VGPR or better rate was defined as the percentage of participants who achieved VGPR or CR (including sCR) according to the IMWG criteria during or after the study treatment. VGPR: Serum and urine component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hour; CR: negative immunofixation on the serum and urine, Disappearance of any soft tissue plasmacytomas and <5% PCs in bone marrow; sCR: CR in addition to having a normal FLC ratio and an absence of clonal cells in bone marrow by immunohistochemistry, immunofluorescence, 2-4 color flow cytometry.
Time Frame: From baseline up to 2 years 7 months
Population: All treated analysis set included all participants who have received at least 1 dose of study treatment. This secondary OM was planned to be analyzed for D-VMP, D-Rd and D-Kd cohorts only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 67 | 65 | 66
percentage of participants | 77.6 [67.6 to 85.7] | 80.0 [70.1 to 87.7] | 77.3 [67.2 to 85.4]

6. Secondary Outcome: D-VRd Cohort: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a PR or better, IMWG criteria, during the study or during follow up. IMWG criteria for PR >= 50% reduction of serum M-protein and reduction in 24 hour urinary M-protein by >=90% or to <200 mg/24 hours, if the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow PCs is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%, in addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Up to 2 years and 3 months
Population: All treated analysis set included all participants who have received at least 1 dose of study treatment. This secondary OM was planned to be analyzed for D-VRd cohort only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd)
Number analyzed (Participants) | 67
percentage of participants | 97.0 [90.9 to 99.5]

7. Secondary Outcome: Percentage of Participants With CR or Better Response
Description: CR or better rate was defined as the percentage of participants with a CR or better response (that is, CR and sCR) as per IMWG criteria. CR: as negative immunofixation on the serum and urine and disappearance of soft tissue plasmacytomas and less than (<) 5 percent plasma cells in bone marrow; sCR: CR plus normal FLC ratio and absence of clonal PCs by immunohistochemistry, immunofluorescence or 2- to 4-color flow cytometry.
Time Frame: For D-VRD Arm: Baseline up to 2 years 3 months; For D-VMP, D-Rd and D-Kd Arms: Baseline up to 2 years 7 months
Population: All treated analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 67 | 67 | 65 | 66
percentage of participants | 16.4 [9.5 to 25.7] | 55.2 [44.5 to 65.6] | 50.8 [39.9 to 61.5] | 42.4 [32.1 to 53.3]

8. Secondary Outcome: D-VMP, D-Rd and D-Kd Cohorts: Duration of Response (DOR)
Description: DOR was defined as the time from the date of initial documented response (PR or better response) to the date of first documented evidence of progressive disease (PD) or death due to PD. PD is defined as an increase of 25% from the lowest response value in one of the following: serum and urine M-component (absolute increase must be >=0.5 gram per deciliter [g/dL] and >=200 mg/24 hours respectively); only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dL); definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From baseline up to 2 years 7 months
Population: Analysis population included number of responders (partial response or better) in each cohort. This secondary outcome measure was planned to be analyzed for D-VMP, D-Rd and D-Kd cohorts.
Measure: Median (Full Range); unit: months
Arm/Group | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 60 | 61 | 56
months | NA [NA to NA] — Here, NA signifies that as per Kaplan-Meier estimate, the median duration of response was not estimable due to less number of events. | NA [NA to NA] — Here, NA signifies that as per Kaplan-Meier estimate, the median duration of response was not estimable due to less number of events. | NA [NA to NA] — Here, NA signifies that as per Kaplan-Meier estimate, the median duration of response was not estimable due to less number of events.

9. Secondary Outcome: Percentage of Participants With Anti-Daratumumab Antibodies
Description: Percentage of participants with antibodies to daratumumab were reported.
Time Frame: For D-VRD Arm: Baseline up to 2 years 3 months; For D-VMP, D-Rd and D-Kd Arms: Baseline up to 2 years 7 months
Population: Immunogenicity-evaluable analysis set was defined as all participants who received at least 1 dose administration of daratumumab SC and had at least 1 immunogenicity sample for detection of anti-daratumumab antibodies after the first dose.
Measure: Number; unit: percentage of participants
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 65 | 64 | 62 | 64
percentage of participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Anti-rHuPH20 Antibodies
Description: Percentage of participants with antibodies to rHuPH20 were reported.
Time Frame: For D-VRD Arm: Baseline up to 2 years 3 months; For D-VMP, D-Rd and D-Kd Arms: Baseline up to 2 years 7 months
Population: Immunogenicity-evaluable analysis set for rHuPH20 is defined as all participants who received at least one dose of daratumumab SC and had appropriate plasma samples for detection of antibodies to rHuPH20 (at least 1 sample after the start of the first dose of daratumumab SC).
Measure: Number; unit: percentage of participants
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 66 | 64 | 62 | 64
percentage of participants | 6.1 | 3.1 | 4.8 | 4.7

11. Secondary Outcome: D-VMP, D-Rd, and D-Kd Cohorts: Percentage of Participants With Minimal Residual Disease (MRD) Negative Rate
Description: MRD negativity rate was defined as the percentage of participants who were considered MRD negative after MRD testing at any timepoint after the first dose by bone marrow aspirate. MRD negativity rate was assessed by next-generation sequencing at a threshold of <10^5.
Time Frame: Up to 2 years and 3 months
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
Number analyzed (Participants) | 67 | 65 | 66
percentage of participants | 25.4 [16.9 to 35.6] | 21.5 [13.5 to 31.6] | 27.3 [18.4 to 37.7]

ADVERSE EVENTS:
Time Frame: For D-VRD Arm: Baseline up to 2 years 3 months; For D-VMP, D-Rd and D-Kd Arms: Baseline up to 2 years 7 months
Description: All treated analysis set included all participants who received at least 1 dose of study treatment.
Arm/Group | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) | D + Bortezomib + Melphalan + Prednisone (D-VMP) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd)
All-Cause Mortality (participants affected / at risk) | 1/67 | 3/67 | 4/65 | 5/66
Serious Adverse Events (participants affected / at risk) | 19/67 | 30/67 | 37/65 | 22/66
Other Adverse Events (participants affected / at risk) | 67/67 | 67/67 | 65/65 | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) (N=67) | D + Bortezomib + Melphalan + Prednisone (D-VMP) (N=67) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) (N=65) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd) (N=66)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 2 | 3 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Ophthalmic Vein Thrombosis (Eye disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 1 | 0
Performance Status Decreased (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 5 | 3 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 2
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Diarrhoea Infectious (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 0
Enterobacter Infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 1 | 0
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 4 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 3 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 6 | 9 | 3
Sepsis (Infections and infestations) | 0 | 0 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 3 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Viral Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0
Body Temperature Increased (Investigations) | 1 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0 | 0 | 0
Respirovirus Test Positive (Investigations) | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 1
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebellar Haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral Small Vessel Ischaemic Disease (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Incoherent (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Thalamic Infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Vith Nerve Paresis (Nervous system disorders) | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2 | 3 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cardiac Ablation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab (D)+Bortezomib+Lenalidomide+Dexamethasone (D-VRd) (N=67) | D + Bortezomib + Melphalan + Prednisone (D-VMP) (N=67) | Daratumumab + Lenalidomide + Dexamethasone (D-Rd) (N=65) | Daratumumab + Carfilzomib + Dexamethasone (D-Kd) (N=66)
Anaemia (Blood and lymphatic system disorders) | 12 | 30 | 26 | 25
Leukopenia (Blood and lymphatic system disorders) | 9 | 8 | 11 | 6
Lymphopenia (Blood and lymphatic system disorders) | 13 | 15 | 10 | 12
Neutropenia (Blood and lymphatic system disorders) | 25 | 30 | 44 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 38 | 23 | 34
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0 | 6
Cataract (Eye disorders) | 0 | 1 | 11 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 4 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 3 | 9 | 3 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 4 | 3 | 4
Constipation (Gastrointestinal disorders) | 26 | 30 | 21 | 6
Diarrhoea (Gastrointestinal disorders) | 16 | 23 | 32 | 20
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 1 | 2
Nausea (Gastrointestinal disorders) | 12 | 23 | 8 | 17
Odynophagia (Gastrointestinal disorders) | 3 | 2 | 2 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 4 | 3 | 0
Vomiting (Gastrointestinal disorders) | 6 | 14 | 7 | 11
Asthenia (General disorders) | 10 | 17 | 21 | 14
Chills (General disorders) | 8 | 3 | 4 | 2
Fatigue (General disorders) | 18 | 10 | 19 | 13
Injection Site Erythema (General disorders) | 9 | 5 | 0 | 5
Malaise (General disorders) | 0 | 5 | 1 | 0
Oedema Peripheral (General disorders) | 13 | 11 | 15 | 12
Pyrexia (General disorders) | 22 | 22 | 16 | 14
Bronchitis (Infections and infestations) | 2 | 17 | 10 | 7
Conjunctivitis (Infections and infestations) | 2 | 5 | 4 | 3
Gastroenteritis (Infections and infestations) | 1 | 7 | 2 | 3
Herpes Zoster (Infections and infestations) | 0 | 6 | 2 | 1
Infection (Infections and infestations) | 0 | 0 | 4 | 3
Nasopharyngitis (Infections and infestations) | 2 | 16 | 8 | 17
Pneumonia (Infections and infestations) | 3 | 6 | 9 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 7 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 19 | 20 | 12
Urinary Tract Infection (Infections and infestations) | 0 | 9 | 8 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 6 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 5 | 4 | 7
Aspartate Aminotransferase Increased (Investigations) | 2 | 4 | 3 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 5 | 3 | 5
Blood Creatinine Increased (Investigations) | 2 | 7 | 8 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 5 | 0 | 8
Weight Decreased (Investigations) | 2 | 7 | 8 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 13 | 4 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 9 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 6 | 9 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 7 | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 4 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 15 | 10 | 13
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 19 | 14 | 11
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 4 | 21 | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 8 | 6 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 11 | 3 | 4
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 6
Dizziness (Nervous system disorders) | 6 | 8 | 9 | 3
Headache (Nervous system disorders) | 7 | 6 | 5 | 15
Paraesthesia (Nervous system disorders) | 2 | 9 | 5 | 6
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 4 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 28 | 26 | 14 | 7
Syncope (Nervous system disorders) | 0 | 4 | 3 | 1
Tremor (Nervous system disorders) | 4 | 3 | 4 | 2
Anxiety (Psychiatric disorders) | 2 | 1 | 4 | 7
Depression (Psychiatric disorders) | 0 | 4 | 4 | 2
Insomnia (Psychiatric disorders) | 12 | 16 | 13 | 23
Irritability (Psychiatric disorders) | 1 | 1 | 2 | 4
Sleep Disorder (Psychiatric disorders) | 0 | 2 | 3 | 4
Acute Kidney Injury (Renal and urinary disorders) | 1 | 3 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 12 | 10 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 16 | 12
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 4 | 7 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 9 | 11 | 10 | 6
Rash Generalised (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 | 4 | 4 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 1 | 4 | 2
Hypertension (Vascular disorders) | 1 | 10 | 8 | 23
Hypotension (Vascular disorders) | 3 | 8 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03412565/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03412565/SAP_003.pdf